CLINICAL TRIAL: NCT00682851
Title: A Validation Study of Genzyme Diagnostics OSOM Trichomonas Rapid Test and BVBlue Test
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sharon Hillier, PhD, University of Pittsburgh
Other Study IDs: PRO08020012
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Results first posted 2011-08-08 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Bacterial Vaginosis; Urogenital Infection by Trichomonas Vaginalis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: OSOM Trichomonas Rapid Test — Rapid test run using vaginal discharge collected via a cotton swab
Device: OSOM BVBlue Test — Rapid test run using vaginal discharge collected using a cotton swab

SUMMARY:
This research is being done to see if two rapid bedside tests (OSOM Trichomonas Rapid Test and BVBlue Test) that give results in 10 minutes are as accurate as standard tests to diagnose common vaginal infections.

DETAILED DESCRIPTION:
This research is being done to see if two rapid bedside tests (OSOM Trichomonas Rapid Test and BVBlue Test) that give results in 10 minutes are as accurate as standard tests (that take up to 7 days to get results) to diagnose common vaginal infections (Trichomonas and bacterial vaginosis).

Both rapid tests (OSOM and BVBlue) are approved by the Food and Drug Administration (FDA) to be used by healthcare professionals to aid in the diagnosis of these infections. This study is being done to validate (or confirm)the accuracy of these tests. This study may help researchers decide if these tests could be used in remote research settings (in place of the standard office testing) to increase diagnosis and prompt treatment of these vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

* At least 15 years of age at time of enrollment
* Ability to provide written informed consent

Exclusion Criteria:

* Currently menstruating or bleeding
* Use of an antibiotic to treat bacterial vaginosis or Trichomonas within the past 7 days

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Non-pregnant women between the ages of 18 and 60, with or without symptoms of vaginitis, were recruited for this study from Magee-Womens Hospital of University of Pittsburgh Medical Center and Allegheny County Health Department.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Symptomatic: Women who presented with one or more symptoms of vaginitis including abnormal vaginal odor, abnormal vaginal discharge, pruritis, vaginal burning or pain, vaginal irritation, or lower abdominal pain.
- Asymptomatic: Women who presented without any symptoms of vaginitis (abnormal vaginal odor, abnormal vaginal discharge, pruritis, vaginal burning or pain, vaginal irritation, or lower abdominal pain).
Period: Overall Study
Arm/Group | Symptomatic | Asymptomatic
Started | 251 | 268
Completed | 251 | 268
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic | Asymptomatic | Total
Number analyzed (Participants) | 251 | 268 | 519
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 16 | 28
  Between 18 and 65 years | 239 | 252 | 491
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (8.2) | 27.0 (8.7) | 27.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 268 | 519
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 251 | 268 | 519

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the OSOM Rapid Test and PCR Wet Mount Microscopy in Diagnosing Trichomonas Vaginalis in Symptomatic and Asymptomatic Women
Description: Sensitivity of the OSOM Rapid test and PCR wet mount microscopy in diagnosing Trichomonas vaginalis using Trichomonas culture as the gold standard in symptomatic and asymptomatic women. The sensitivity of a test is the percentage of people who have the infection (as diagnosed by the gold standard method) among those who have a positive test.
Time Frame: Visit 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 251 | 268
Percentage of Participants
  OSOM Rapid Test | 92 [78 to 98] | 91 [72 to 99]
  PCR | 100 [90 to 100] | 100 [85 to 100]
  Wet Mount Microscopy | 58 [41 to 74] | 48 [27 to 69]

2. Secondary Outcome: Specificity of the OSOM Rapid Test and PCR Wet Mount Microscopy in Diagnosing Trichomonas Vaginalis in Symptomatic and Asymptomatic Women
Description: Specificity of the OSOM Rapid test and PCR wet mount microscopy in diagnosing Trichomonas vaginalis using Trichomonas culture as the gold standard in symptomatic and asymptomatic women. The specificity of a test is the percentage of people who do not have the infection (as diagnosed using the gold standard method) among those who have a negative test.
Time Frame: Visit 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 251 | 268
Percentage of Participants
  OSOM Rapid Test | 99 [97 to 100] | 99 [97 to 100]
  PCR | 96 [92 to 98] | 96 [92 to 98]
  Wet Mount Microscopy | 99 [97 to 100] | 100 [99 to 100]

3. Secondary Outcome: Sensitivity of the BVBlue Test and Amsel Criteria in Diagnosing Bacterial Vaginosis in Symptomatic and Asymptomatic Women.
Description: Sensitivity of the BVBlue Test and Amsel criteria in diagnosing bacterial vaginosis using Gram Stain (Nugent scoring) as the gold standard in symptomatic and asymptomatic women. The sensitivity of a test is the percentage of people who have the infection (as diagnosed by the gold standard method) among those who have a positive test.
Time Frame: Visit 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 251 | 268
Percentage of Participants
  BVBlue Test | 68 [60 to 76] | 61 [51 to 71]
  Amsel Criteria | 82 [75 to 88] | 67 [57 to 76]

4. Secondary Outcome: Specificity of the BVBlue Test and Amsel Criteria in Diagnosing BV in Symptomatic and Asymptomatic Women.
Description: Specificity of the BVBlue Test and Amsel criteria in diagnosing BV using Gram Stain (Nugent scoring) as the gold standard in symptomatic and asymptomatic women. The specificity of a test is the percentage of people who do not have the infection (as diagnosed by the gold standard method) among those who have a negative test.
Time Frame: Visit 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 251 | 268
Percentage of Participants
  BVBlue Test | 100 [96 to 100] | 99 [96 to 100]
  Amsel Criteria | 94 [87 to 98] | 100 [98 to 100]

ADVERSE EVENTS:
Arm/Group | Symptomatic | Asymptomatic
Serious Adverse Events (participants affected / at risk) | 0/251 | 0/268
Other Adverse Events (participants affected / at risk) | 0/251 | 0/268

LIMITATIONS AND CAVEATS:
A major limitation of this study was that in the first 122 women, 24% of the cohort, the vaginal swabs used for the diagnostic tests were collected in random order, which resulted in decreased sensitivity of the OSOM Rapid and BVBLue tests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No